CLINICAL TRIAL: NCT04430166
Title: A Exploratory Clinical Study on PD-1 Monoclonal Antibody in Pre-treated Lymphoepithelioma-like Carcinoma
Brief Title: PD-1 Monoclonal Antibody in Pre-treated Lymphoepithelioma-like Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Haibo Zhang, Professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019KT1192
Record Dates: First submitted 2020-05-28; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2019-12

CONDITIONS: Lymphoepithelioma-Like Carcinoma
Keywords: Lymphoepithelioma-like carcinoma; PD-1 monoclonal antibody
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 monoclonal antibody (Experimental)
  Interventions: Drug: PD-1 monoclonal antibody

INTERVENTIONS:
Drug: PD-1 monoclonal antibody — 200mg / intravenous drip, once every three weeks

SUMMARY:
Lymphoepithelioma-like carcinoma (LELC) may benefit from immunocheckpoint inhibitor therapy. Although target antibody drugs for PD-1 and PD-L1 have achieved good results in immunotherapy of many malignant tumors, there is still a lack of corresponding clinical research reports on whether LELC treatment can benefit. Therefore, this study intends to adopt the basket research model , to explore the application of anti-procedural death receptor 1 (PD-1) monoclonal antibody in patients with advanced LELC after the failure of first-line standard treatment . Further explore the relationship between tumor and body immunity, tumor microenvironment and curative effect, and find stable biomarkers, so as to screen out the superior population of tumor immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of lymphoepithelioma-like carcinoma
* Failed the first-line standard treatment or progressed after the treatment, at least one measurable lesion according to the RECIST1.1 standard
* Age between 18 and 80 years old
* Estimated life expectancy exceeds 3 months
* ECOG Performance Status score ≤ 2
* Normal bone marrow, liver, kidney, clotting function, including： hemoglobin ≥90g/L (no history of blood transfusion within 7 days), absolute neutrophil count ≥1.5×109/L, platelet ≥100×109/L, total bilirubin ≤1.5×ULN, albumin ≥30g/ L, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN), if combined with liver metastases, AST and ALT ≤ 5 × ULN; creatinine ≤ 1.5 × ULN; international standardized ratio (INR) or coagulation Proenzyme time (PT) ≤ 1.5 × ULN, if the subject receives anticoagulant therapy normally, as long as the PT is within the range planned by the anticoagulant drug
* Women of childbearing age should have a urine or serum pregnancy test negative within 3 days before receiving the first study drug administration. If the urine pregnancy test result cannot be confirmed negative, a blood pregnancy test is required
* Ensure effective contraception during the study period and at least 6 months after the study ended.
* Sign an informed consent form and follow up with good compliance

Exclusion Criteria:

* Merging other pathological tumors
* Active bleeding, active diverticulitis, abdominal abscess, gastrointestinal perforation, gastrointestinal obstruction, and peritoneal metastasis that require clinical intervention; clinically uncontrollable pleural, abdominal, and pericardial effusions (drainage effusions are not required or patients who have stopped draining for 3 days without a significant increase in effusion can be enrolled); severe bleeding tendency or coagulopathy；receiving thrombolytic therap
* Uncontrolled hypertension（systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg after optimal medical treatment）；history of hypertension crisis or hypertensive encephalopathy
* History of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation)
* Grade III-IV congestive heart failure (according to New York Heart Association classification), poorly controlled and clinically significant
* Any arterial, venous thrombosis, embolism, or ischemia occurred within 6 months before enrolling in the treatment
* Central nervous system metastasis
* Active infection that requires treatment, or systemic anti-infective drugs have been used within one week before the first dose; or there is active tuberculosis (TB), normal anti-TB treatment or anti-TB within 1 year before the first dose treatment
* Known history of human immunodeficiency virus (HIV) infection (ie HIV1/2 antibody positive), known syphilis infection
* Acute or chronic active hepatitis B or hepatitis C infection, including hepatitis B virus (HBV) DNA>2000IU/ml or 104 copies/ml，hepatitis C virus (HCV) RNA>103 copies/ml or HBsAg Positive simultaneously with anti-HCV antibody
* Active autoimmune diseases requiring systemic treatment occurred within 2 years before the first dose(alternative therapies such as thyroxine, insulin, or physiological doses of corticosteroids used for adrenal or pituitary insufficiency are not considered systemic treatment）
* History of non-infectious pneumonia requiring corticosteroid therapy or current pneumonia within 1 year before the first dose（patients with intermittent use of bronchodilators, inhaled corticosteroids, or local injection of corticosteroids due to COPD and asthma can be enrolled）
* Previously received immunotherapy treatment, or received immunomodulatory drug treatment within 2 weeks before the first dose, or received major surgical treatment within 3 weeks before the first dose
* Known to have an allergic reaction to the active ingredient of PD-1 monoclonal antibody and/or any excipients
* Mental illnesses or drug abuse that may affect compliance with research requirements
* Currently participating in interventional clinical research treatment, or receiving other research drugs or research equipment within 4 weeks before the first dose
* Women who are pregnant or breastfeeding
* Other acute, chronic and mental diseases that may lead to the following results: laboratory test values are abnormal；increase the risk of research participation or study drug administration； interfere with the interpretation of the study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | Through study completion, an average of 9 weeks
  The time from enrollment to the occurrence of tumor development (in any aspect) or death (for any reason).
  For subjects without disease progression or death, the date of the last imaging evaluation is the date of censorship. Subjects who did not undergo imaging evaluation or no death record after baseline were deleted based on the enrollment date.

SECONDARY OUTCOMES:
Objective response rate | Through study completion，an average of 9 weeks
  According to the RECIST 1.1 standard, the proportion of subjects with complete response(CR) or partial response(PR) in the analysis population.
Time to initial response | Through study completion，an average of 9 weeks
  The time from enrollment to the first objective response (CR or PR) of the tumor.
  For subjects who did not reach CR or PR, the date of the last imaging evaluation was the date of censorship.
Overall survival | Through study completion， an average of 90 days
  The time from enrollment to (for any reason) death. At the end of the study, if the subject is still alive, the known date of the subject's last survival" will be the censored date.
Duration of response | Through study completion，an average of 9 weeks
  The time from the first recorded objective tumor response (CR or PR) to objective disease progression (PD) or death.
  For subjects without disease progression or death, the date of the last imaging evaluation is the date of censorship.
Tumor immune microenvironment | Baseline
  immune microenvironment state of tumor tissue will be detected by Opal multiplex immunofluorescence assay

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No